CLINICAL TRIAL: NCT02726191
Title: Computerized Cognitive Training in Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Lapsed
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-00398
Record Dates: First submitted 2016-03-22; First posted 2016-04-01 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posit Science (Experimental)
  Interventions: Behavioral: Spatial Match Exercise; Behavioral: Temporal Sequence Reconstruction Exercise; Behavioral: Token Task Exercise; Behavioral: Story Recall Exercise; Behavioral: Sample-Match (Within Modality) Exercise; Behavioral: Pair-Match (Across-Modality) Exercise; Behavioral: Triad-FiguresExercise
- Lumosity (Experimental)
  Interventions: Behavioral: Monster Garden Exercise; Behavioral: Memory Match Exercise; Behavioral: Memory Matrix Exercise; Behavioral: Familiar Faces Exercises; Behavioral: Lost in Migration Exercise; Behavioral: Playing Koi Exercise

INTERVENTIONS:
Behavioral: Spatial Match Exercise
  Arms: Posit Science
Behavioral: Temporal Sequence Reconstruction Exercise
  Arms: Posit Science
Behavioral: Token Task Exercise
  Arms: Posit Science
Behavioral: Story Recall Exercise
  Arms: Posit Science
Behavioral: Sample-Match (Within Modality) Exercise
  Arms: Posit Science
Behavioral: Pair-Match (Across-Modality) Exercise
  Arms: Posit Science
Behavioral: Triad-FiguresExercise
  Arms: Posit Science
Behavioral: Monster Garden Exercise
  Arms: Lumosity
Behavioral: Memory Match Exercise
  Arms: Lumosity
Behavioral: Memory Matrix Exercise
  Arms: Lumosity
Behavioral: Familiar Faces Exercises
  Arms: Lumosity
Behavioral: Lost in Migration Exercise
  Arms: Lumosity
Behavioral: Playing Koi Exercise
  Arms: Lumosity

SUMMARY:
The purpose of this randomized uncontrolled single-site trial is to evaluate the efficacy of two novel computerized cognitive enhancing software packages for improving cognitive and behavioral outcomes in patients with epilepsy.

DETAILED DESCRIPTION:
The proposed investigation will be the first to pit two software packages against each other to evaluate the relative efficacy and feasibility of their use among patients with epilepsy. Pharmacotherapy fails to control seizures in approximately 30% of patients. Use of non-pharmacologic interventions, such as cognitive rehabilitation, has shown some benefit for improving cognitive functions and reducing mood symptoms. Each of the computer exercises employ a set of stimuli that are generalizable and mimic real-world experiences.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of epilepsy based on medical records. The records will be reviewed by the PI and the approved study personnel to confirm that a diagnosis of epilepsy has been made.
* Must own a computer or have access to the internet.

Exclusion Criteria:

* Full Scale IQ < 80, as assessed by the WASI-II.
* History of chronic progressive neurologic or neurodegenerative illnesses (e.g., Parkinson's disease, multiple sclerosis, dementia, primary or metastatic malignancy). Patients with headache or migraine are not excluded.
* History of Axis I psychiatric illness with psychotic features. (e.g., schizophrenia). Patients with depression or anxiety (treated or untreated) without psychotic features are not excluded.
* Visual or auditory impairment, which precludes participation in part, or all of the testing.
* English as a first language will not be required, but participants must have either received some of their schooling in English or used English in their work for >10 years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-07 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Total Index Score from the Repeatable Battery for the Assessment of Neurocognitive Status (RBANS) | 8 Weeks

SECONDARY OUTCOMES:
The Everyday Cognition Scale (ECog) | 8 Weeks
Perceived cognitive abilities on an index of subjective cognitive abilities (Cognitive Self-Report Questionnaire; CSRQ-25) | 8 Weeks
Measure of mood (Geriatric Depression Scale) | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stella Karantzoulis, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States